CLINICAL TRIAL: NCT04602936
Title: Solriamfetol in Binge Eating Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lindner Center of HOPE (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Jazz BED
Record Dates: First submitted 2020-10-14; First posted 2020-10-26 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Binge Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — solriamfetol

STUDY DESIGN:
Intervention Model Description: This is a 1-site, randomized, parallel group, double-blind, placebo-controlled, flexible-dose study in which solriamfetol 37.5-150 mg/day will be administered for 12 weeks to 64 outpatient adults with BED by DSM-5 criteria
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Solriamfetol (Active Comparator): All medication will be 37.5 mg encapsulated soriamfetol tablets or matching encapsulated placebo tablets supplied in numbered containers for dispensing to patients. The minimum dose of solriamfetol during the trial will be 37.5 mg/day; the maximum dose will be 150 mg/day. At the Baseline Visit (Visit 0), participants will be instructed to take one capsule of solriamfetol 37.5 mg or matching placebo in the morning for the first 7 days. Thereafter, at Visit 1, solriamfetol or placebo will be increased to 75 mg/day, if tolerated. Beginning on day 15 (Visit 2), solriamfetol or placebo will be increased to 150 mg/day, if tolerated. Study medication dosage may be decreased, or a scheduled increase may not be made, because of side effects. Study medication will be administered as a single daily dose in the morning.
  Interventions: Drug: Solriamfetol
- Placebo (Placebo Comparator): Placebo (i.e., inactive compound for comparison)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Solriamfetol — Solriamfetol is a novel DNRI (novel dopamine and norepinephrine reuptake inhibitor) that has recently received regulatory approval for the treatment of excessive daytime sleepiness in individuals with narcolepsy or obstructive sleep apnea.
  Other Names: Sunosi
  Arms: Solriamfetol
Drug: Placebo — A placebo is a substance or treatment which is designed to have no therapeutic value (an inactive compound, i.e. inert, often called a "sugar pill").
  Arms: Placebo

SUMMARY:
The goal of this project is to evaluate the efficacy and tolerability of the novel dopamine and norepinephrine reuptake inhibitor (DNRI) solriamfetol in the treatment of binge eating disorder (BED).

DETAILED DESCRIPTION:
This is a 1-site, randomized, parallel group, double-blind, placebo-controlled, flexible-dose study in which solriamfetol 37.5-150 mg/day will be administered for 12 weeks to 64 outpatient adults with BED by DSM-5 criteria. The study will have 3 phases: a 1-2 week Screening phase to evaluate participant eligibility; a 12-week blinded Treatment phase during which participants will receive solriamfetol or matching placebo; and a 1-week Treatment Discontinuation phase. During the Treatment phase, participants will be evaluated weekly for the first 4 weeks and then biweekly for the next 8 weeks. Solriamfetol will be started at 37.5 mg/day. After 1 week, study drug will be increased to 75 mg/day. If a participant continues to have BED symptoms, study drug may be increased to a maximum of 150 mg/d by Treatment week 6; after that, study drug dose will be held constant. Efficacy will be assessed by measuring the weekly frequency of binge-eating episode days with patient take-home diaries. Regular monitoring of vital signs, laboratory tests, electrocardiograms (ECGs), adverse events, and suicidality will assess safety

ELIGIBILITY:
Inclusion Criteria: Criteria for entering this study will include all of the following:

1. Participants will meet DSM-5 criteria for a diagnosis of BED. These criteria are:

   1. Recurrent episodes of binge eating. Both of the following characterize a binge-eating episode: 1. Eating, in a discrete period (e.g., within 2 hours), an amount of food that is definitely larger than most people would eat in a similar period under similar conditions; and 2. A sense of lack of control over the eating (e.g., a feeling that one cannot stop eating or control what or how much one is eating).
   2. The binge-eating episodes are associated with at least three of the following: eating much more rapidly than normal; eating until uncomfortably full; eating large amounts of food when not feeling physically hungry; eating alone because of being embarrassed by how much one is eating; feeling disgusted with oneself, depressed, or feeling very guilty after overeating.
   3. Marked distress regarding binge eating.
   4. The binge eating occurs, on average, at least one day a week for 3 months.
   5. The episodes of binge eating do not occur exclusively during the course of bulimia nervosa or anorexia nervosa.
2. In addition, to ensure that BED is of at least moderate severity, participants will report at least three binge-eating days per week during the 1 week prior to initiation of study medication, prospectively documented in take-home binge diaries. A binge-eating day (or binge day) is a day during which at least one binge-eating episode occurs.
3. Men or women, through the ages of 18 and 65 years, inclusive.

Exclusion Criteria: Criteria for exclusion from this study will be any of the following:

1. Have a current diagnosis of bulimia nervosa or anorexia nervosa.
2. Women who are pregnant, lactating, or of childbearing potential who are not using adequate contraceptive measures. The following are considered adequate methods of birth control: 1. intrauterine device (IUD); 2. barrier protection; 3. a contraceptive implantation system (Norplant); 4. oral contraceptive pills; 5. a surgically sterile patient; and 6. abstinence. All female participants will have a negative pregnancy test prior to randomization.
3. Individuals who are displaying clinically significant suicidality or homicidality.
4. Individuals who are receiving a psychological (e.g., supportive psychotherapy, cognitive behavior therapy, interpersonal therapy) or weight loss (e.g., Weight Watchers) intervention for BED that was begun within the 3 months before study entry. Individuals beginning such treatment more than 3 months prior to study entry may be enrolled as long as they to agree to not make any changes to the frequency or nature of their treatment during the course of the drug trial.
5. A DSM-IV-TR diagnosis of substance abuse or dependence (except nicotine abuse or dependence) within the 6 months prior to randomization.
6. Individuals who have used psychostimulants to facilitate fasting or dieting as a part of their eating disorder within the past 6 months, individuals who have misused psychostimulants within the past 6 months, and individuals who have a drug screen at the Screening visit positive for psychostimulants.
7. Individuals with a lifetime DSM-IV-TR history of psychosis, mania or hypomania, or dementia.
8. Individuals with a history of any psychiatric disorder that might interfere with a diagnostic assessment, treatment, or study compliance.
9. Individuals who have a body mass index (BMI) ≤ 18 mg/kg2
10. Clinically unstable medical disease, including cardiovascular, hepatic, renal, gastrointestinal, pulmonary, metabolic, endocrine, or other systemic disease.
11. Have a history of a structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormality, coronary artery disease, stroke, or other serious cardiovascular problem.
12. History of seizures, including clinically febrile seizures in childhood.
13. Have uncontrolled hypertension (>160/100) or tachycardia (heart rate >110).
14. Have an ECG with significant arrhythmias or conduction abnormalities, which in the opinion of the physician investigator precludes study participation.
15. Have clinically relevant abnormal laboratory results, specifically including hypokalemia.
16. Have a history of narcolepsy or obstructive sleep apnea, or currently receiving treatment with an alerting agent.
17. Individuals requiring treatment with any drug which might interact adversely with or obscure the action of the study medication. This includes warfarin, anticonvulsants, clonidine, theophylline, and pseudoephedrine.
18. Individuals who have received any psychotropic medications (other than hypnotics) within four weeks prior to randomization, including antidepressants (including monoamine oxidase inhibitors), antipsychotics, mood stabilizers, or psychostimulants.
19. Individuals who have received investigational medications or depot neuroleptics within three months prior to randomization.
20. Individuals who have a known allergy to solriamfetol or its constituents.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy variable is binge-eating day frequency as assessed by the take-home patient diary. | Days 1-84
  days with binge eating episodes

SECONDARY OUTCOMES:
The secondary efficacy variables will include binge-eating episode frequency. | Days 1-84
  Number of binge eating episodes per week
The score on the Yale-Brown Obsessive Compulsive Scale Modified for Binge Eating (YBOC-BE). | Weeks 1, 2, 3, 4, 6, 8, 10, 12
  Questions on scale range from 0-4, higher scores are worse. There are 10 questions total. The first 5 questions consist of the "obsessional sub-total" (scores are added together). Questions 6-10 are added together and equal the "compulsion sub-total."
The score on the Clinical Global Impression-Severity (CGI-S) and Clinical Global Impressions-Improvement scale (CGI-I). | Weeks 1, 2, 3, 4, 6, 8, 10, 12
  The Clinical Global Impression - Severity and Improvement scale (CGI-S, CGI-I) is a 7-point scale that requires the clinician to rate the severity and improvement of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. On the CGI-S question, scores range from 1-7, with higher scores being worse (1 = normal, 7 = very severely ill). On the CGI-I questions, scores range from 1-8, with higher scores being worse (1 = no change, 7 = very much worse, 8 = not applicable).

CONTACTS AND LOCATIONS:
Locations (1):
- Lindner Center of HOPE, Mason, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guerdjikova AI, Romo-Nava F, Blom TJ, Mori N, McElroy SL. Study protocol and rationale for a randomized, placebo-controlled trial of solriamfetol to treat binge eating disorder. Contemp Clin Trials. 2021 Nov;110:106587. doi: 10.1016/j.cct.2021.106587. Epub 2021 Oct 2. PMID 34610482